CLINICAL TRIAL: NCT01159236
Title: Molecular Triaging of Newly Diagnosed Breast Cancer for Preoperative Therapies
Brief Title: Molecular Triaging of Newly Diagnosed Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recent developments lead to re-evaluation of study.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0765
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Gene signatures; HER-2 normal stage I-III breast cancer; Estrogen Receptor; ER-positive; ER-negative; RCB categories II-III; Neoadjuvant Chemotherapy; adjuvant systemic therapy; molecular testing; Fluorouracil; 5-fluorouracil; 5-FU; Doxorubicin; Adriamycin; Rubex; Epirubicin; Ellence; Cyclophosphamide; Cytoxan; Neosar; Bevacizumab; Avastin; Anti-VEGF monoclonal; rhu-MAb-VEGF
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Fluorouracil; Doxorubicin; Epirubicin; Cyclophosphamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: ER-Positive (Experimental): Participants with Estrogen Receptor (ER)-Positive breast cancers receive Standard T/FAC or T/FEC chemotherapy before surgery.
  T/FAC or T/FEC: Combination chemotherapy with sequential paclitaxel (80 mg/m2) weekly x 12 weeks followed by 5-fluorouracil (500 mg/m2), cyclophosphamide (500 mg/m2) and doxorubicin (50 mg/m2) or epirubicin (100 mg/m2) (FAC or FEC) once every 3 weeks for 4 treatments.
  Interventions: Drug: Paclitaxel; Drug: Fluorouracil; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide
- Group 2: ER-Negative (Experimental): Participants with ER-negative cancers (randomized between Group 2 & Group 3), Standard T/FAC or T/FEC chemotherapy before surgery.
  Interventions: Drug: Paclitaxel; Drug: Fluorouracil; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide
- Group 3: ER-Negative + Bevacizumab (Experimental): Participants with ER-negative cancers (randomized between Group 2 & Group 3), T/FEC chemotherapy combined with 10 mg Bevacizumab every 2 weeks during first 3 treatments before surgery.
  Interventions: Drug: Paclitaxel; Drug: Fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 by vein over about 1-2 hours once every 7 days x 12 courses.
  Other Names: Taxol
Drug: Fluorouracil — 500 mg/m2 for 4 courses (once every 7 days)
  Other Names: 5-FU; Adrucil; Efudex
Drug: Doxorubicin — 50 mg/m2 by vein given on day 1 and repeated once every 21 days for 4 treatments
  Other Names: Rubex; Adriamycin
  Arms: Group 1: ER-Positive; Group 2: ER-Negative
Drug: Epirubicin — 100 mg/m2 by vein given on day 1 and repeated once every 21 days for 4 treatments, may be given instead of Doxorubicin in Group 1 and 2.
  Other Names: Ellence
Drug: Cyclophosphamide — 500 mg/m2 by vein given on day 1 and repeated once every 21 days for 4 treatments.
  Other Names: Cytoxan; Neosar
Drug: Bevacizumab — 10 mg/kg intravenously every 2 weeks, discontinued 6 weeks before surgery (i.e. after 3rd course of FEC or FAC)
  Other Names: Avastin; Anti-VEGF monoclonal; rhuMAb-VEGF
  Arms: Group 3: ER-Negative + Bevacizumab

SUMMARY:
The goal of this clinical research study is to learn if using "gene signatures" can be an effective way to decide the best treatment for breast cancer patients. Gene signatures may be able to help researchers predict who will respond to chemotherapy given before surgery.

DETAILED DESCRIPTION:
At this time, treatment of stage I-III breast cancer for patients who are at high risk for the cancer returning is surgery and chemotherapy. If the cancer is positive for estrogen hormone receptor, patients also have endocrine therapy.

The most common standard chemotherapy treatment regimens for breast cancer at M. D. Anderson are paclitaxel (T), followed by treatments with fluorouracil (F), doxorubicin (A) or epirubicin (E), and cyclophosphamide (C). These chemotherapy combinations are known as T/FAC and T/FEC. However, not all patients respond to these treatments, so researchers at M. D. Anderson have developed tests to predict how much a person's breast cancer might respond to T/FAC or T/FEC chemotherapy.

Fine needle aspiration (FNA) of the tumor are collected after numbing the skin of the breast with local anesthesia, and the genes within the FNA sample are measured to calculate the results of treatment prediction tests before treatment is selected.

In this research study, the gene-based tests will help to select treatment based on the predictions of response to chemotherapy, and to then measure the tumor response from the surgery after the treatment.

Study Drugs:

T/FAC and T/FEC are designed to damage the DNA (genetic material of cells), which may cause cancer cells to die.

Bevacizumab is designed to block the growth of blood vessels that supply nutrients necessary for tumor growth. This may prevent or slow down the growth of cancer cells and make them more susceptible to chemotherapy.

Tumor Biopsies:

If you are found eligible to take part in this study, you will have 3-4 fine needle biopsies of the tumor collected. The skin over the tumor and the breast tissues surrounding the tumor will be numbed using local anesthesia. To perform fine needle aspiration biopsies, tumor cells are withdrawn from the tumor using a very thin needle alone, or using a syringe.

These biopsies will be used to measure different genes and to predict how the cancer may respond to different treatments.

Based on the information from these gene measurements, a computer model will predict if the cancer is highly sensitive to chemotherapy and is likely to shrink to a great extent or disappear completely due to chemotherapy. This response prediction is done separately for estrogen receptor-positive and estrogen receptor-negative cancers.

Study Groups:

If the biopsies show that the cancer may respond well to standard T/FAC or T/FEC chemotherapy, you will receive the chemotherapy before surgery (Group 1).

If the biopsies show that the cancer may not respond as well to standard T/FAC or T/FEC chemotherapy, you will be randomly assigned (as in the roll of dice) to 1 of 2 groups.

* If you are in Group 2, you will receive T/FAC or T/FEC chemotherapy before surgery. One (1) out of 3 participants whose cancer may not respond as well will be assigned to this group.
* If you are in Group 3, you will receive T/FAC or T/FEC chemotherapy combined with bevacizumab before surgery. Two (2) out of 3 participants whose cancer may not respond as well will be assigned to this group.

Your doctor will decide if you receive T/FAC or T/FEC.

Study Drug Administration:

Groups 1 and 2:

Once a week during Weeks 1-12, you will receive paclitaxel by vein over about 1-2 hours.

Once every 3 weeks during Weeks 13-24, you will receive T/FAC or T/FEC by vein over about 3-4 hours. This chemotherapy treatment is considered routine standard of care and you may receive this treatment closer to home outside of M. D. Anderson.

After all chemotherapy, you will have surgery at M. D. Anderson to remove the cancer.

Group 3:

Once a week during Weeks 1-12, you will receive paclitaxel by vein over about 1-2 hours.

Once every 2 weeks during Weeks 1-18, you will receive bevacizumab by vein once over about 1-2 hours. If your doctor thinks is it necessary, and based on heart related test results, you may only receive bevacizumab during Weeks 1-12.

Once every 3 weeks during Weeks 13-24, you will receive T/FAC or T/FEC by vein over about 4 hours. You must receive your chemotherapy at M. D. Anderson if you are in this group.

After all chemotherapy, you will have surgery at M. D. Anderson to remove the cancer.

Study Visits:

All participants will have routine visits at M. D. Anderson at least once every 12 weeks during chemotherapy. Your doctor will determine the tests and procedures to be performed.

If you are assigned to Group 3, you will also have the following additional procedures.

* You will have a urine analysis within 1 month after starting therapy.
* You will have an echocardiogram to check your heart's health within 3 months after you begin treatment.

Length of Study:

You may receive chemotherapy for up to 6 months. Once surgery is performed, your participation in this study is complete. Your doctor will decide together with you what further treatment you will need after surgery.

This is an investigational study. The biopsy and testing to predict response to chemotherapy is not FDA approved or commercially available. Its use in this study is investigational. The chemotherapy and surgery are standard of care for patients with breast cancer. The addition of bevacizumab to treatment is also investigational.

Up to 303 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older with histologically confirmed HER2-normal (defined as fluorescence in situ hybridization, FISH < 2.2 or immunohistochemistry, IHC <3+ if FISH result is not available) invasive carcinoma of the breast for whom systemic adjuvant therapy is clinically indicated.
2. Patients must have intact cancer in the breast and intact regional lymph nodes (diagnostic core needle or fine needle biopsies are allowed).
3. Routine estrogen, progesterone and HER-2 receptor determination must be performed before starting therapy.
4. Patients with prior history of breast cancer are eligible.
5. Patients with bilateral breast cancers are eligible.
6. Women of childbearing potential must have a negative serum pregnancy test within 2 weeks of starting chemotherapy. Patients must agree to barrier contraception (condom) while on study.
7. Patients must agree to undergo pretreatment needle biopsy of the primary tumor in the breast for molecular profiling.
8. Patients must agree to undergo surgery at MDACC and if assigned to bevacizumab containing chemotherapy it must be administered at MDACC.

Exclusion Criteria:

1. Patients for whom anthracycline or paclitaxel chemotherapies are contraindicated, including: uncompensated congestive heart failure, myocardial infarction within the past 12 months, pre-existing peripheral neuropathy > grade 2, prior doxorubicin therapy with > cumulative dose of 240 mg/m^2
2. Women who had lumpectomy or surgical partial excisional biopsy of the cancer, or sentinel lymph node biopsy of a positive node, before starting preoperative therapy.
3. Exclusion criteria for bevacizumab therapy; inadequately controlled hypertension (defined as systolic blood pressure >/= 140 mmHg and/or diastolic blood pressure >/= 90 mmHg).
4. Exclusion criteria for bevacizumab therapy, prior history of hypertensive crisis or hypertensive encephalopathy, stroke or transient ischemic attacks.
5. Exclusion criteria for bevacizumab therapy, history of myocardial infarction, unstable angina or congestive heart failure within 12 months prior to starting therapy.
6. Exclusion criteria for bevacizumab therapy, aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis within 6 months prior to starting therapy.
7. Exclusion criteria for bevacizumab therapy, history of hemoptysis ( 1/2 teaspoon of bright red blood per episode) within 1 month prior to starting therapy or evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
8. Exclusion criteria for bevacizumab therapy. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting therapy or core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to starting therapy.
9. Exclusion criteria for bevacizumab therapy, history of abdominal fistula or gastrointestinal perforation within 6 months prior to starting therapy.
10. Exclusion criteria for bevacizumab therapy, serious, non-healing wound or fracture or active ulcer.
11. Proteinuria within 1 months of starting therapy as demonstrated by either (a) Urine protein:creatinine (UPC) ratio >/= 1.0 or (b) proteinuria >/= 2+ by urine dipstick test. Patients discovered to have >/=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09

PRIMARY OUTCOMES:
Pathological Response Rate in Patients | Every 3-4 weeks during chemotherapy.
  Response is defined as pathologic complete (pCR/RCB-0) or near complete (RCB-I) response pathologic finding after completion of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, DPHIL, Study Chair — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org